CLINICAL TRIAL: NCT02999919
Title: The Relationship Between Body Mass Index and Post-dural Puncture Headache in Pregnant Women
Brief Title: Body Mass Index and Post-dural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Serbülent Gökhan BEYAZ, associate professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 16214662/050.01.04/87
Record Dates: First submitted 2016-12-18; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: This Study Investigated the Influence of Body Mass Index (BMI) on PDPH in Elective Caesarean Section Patients in Whom 27G Spinal Needles Were Used
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMI ≥ 30 (Active Comparator): BMI ≥ 30
  Interventions: Procedure: spinal anesthesia
- BMI < 30 (Active Comparator): BMI <30
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — 12.5 mg hyperbaric bupivacaine intrathecally following a successful dural puncture performed with a 27G Quincke spinal needle at the L3-4 or L4-5 intervertebral space in the sitting position
  Other Names: bupivacaine

SUMMARY:
Post-dural puncture headache (PDPH) is seen more frequently in pregnant women due to stress, dehydration, intra-abdominal pressure, and insufficient fluid replacement after delivery. Obesity protects against PDPH in pregnant women; increased intra-abdominal fat tissue reduced cerebrospinal fluid leakage by increasing the pressure in the epidural space. Therefore, this study investigated the influence of body mass index (BMI) on PDPH in elective caesarean section patients in whom 27G spinal needles were used.

DETAILED DESCRIPTION:
The study included 420 women with American Society of Anesthesiology physical status I-II who underwent elective caesarean section under spinal anesthesia. The patients with a BMI less than 30 were accepted as normal weight (Group I) and those with a BMI above 30 were accepted as obese (Group II). Dural puncture performed with a 27G Quincke spinal needle at the L3-4 or L4-5 intervertebral space and given 12.5 mg hyperbaric bupivacaine intrathecally. The patients were questioned regarding headache and low back pain 6, 12, 24, and 48 hours after the procedure, and by phone calls on days 3 and 7.

ELIGIBILITY:
Inclusion Criteria:

(ASA) physical status I-II who underwent elective caesarean section under SA. Women age 18-40 years.

Exclusion Criteria:

* Who had undergone lumbar disc or vertebra surgery, had chronic low back pain or headache, had contraindications for neuro-axial block, and emergency patients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
influence of body mass index (BMI) on PDPH in elective caesarean section patients | one year

IPD SHARING:
Plan to Share IPD: No